CLINICAL TRIAL: NCT00743353
Title: An Exploratory, Multi-Center, Open Label, Non-Randomized Study of F-18 RGD-K5
Brief Title: Exploratory, Phase 0 Study of Positron Emission Tomography (PET) Imaging Agent, F-18 RGD-K5
Acronym: K5
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Siemens Molecular Imaging (Industry)
Responsible Party: James Zhang, MD, PhD, MBA, Senior Director, Medical Monitor, Global Head of Clinical Development
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: K5-100
Record Dates: First submitted 2008-08-26; First posted 2008-08-28 (Estimated); Last update posted 2009-02-02 (Estimated); Status verified 2009-01

CONDITIONS: Sarcoma; Melanoma; Lung Cancer; Breast Cancer; High Grade Gliomas
Keywords: laryngeal; squamous cell; anaplastic astrocytoma; oligodendroglioma; glioblastoma multiforme
MeSH Terms: conditions — Sarcoma; Melanoma; Lung Neoplasms; Breast Neoplasms; Laryngeal Diseases; Astrocytoma; Oligodendroglioma; Glioblastoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- A (Experimental): 16 subjects to be enrolled; Study Drug F-18 RGD-K5 administered for diagnostic PET Imaging to be observed for a maximum of 4 hours, followed by 24 hour follow up
  Interventions: Drug: F-18 RGD-K5

INTERVENTIONS:
Drug: F-18 RGD-K5 — Study Drug F-18 RGD-K5 administered for diagnostic PET Imaging to be observed for a maximum of 4 hours, followed by 24 hour follow up

SUMMARY:
The purpose of this research study is to get information from volunteers without cancer and patients with cancer who have received a new investigational study agent called, "[F-18] RGDK5," to evaluate biodistribution and dosimetry for the study agent and determine F-18 RGD-K5 uptake in angiogenic tumor. the system.

DETAILED DESCRIPTION:
[F-18]RGD-K5 is being investigated as a diagnostic radiopharmaceutical for the detection and localization of angiogenesis tissue or lesions supporting the application and role of integrins in anti-angiogenic therapies to benefit patients with cancer and inflammatory diseases.

The primary objectives of this exploratory study are:

* To gain information on biodistribution of [F-18]RGD-K5, and to evaluate the PET images with [F-18]RGD-K5 for resolution, signal to background ratio and for the detection and localization of angiogenesis tissue. This Exploratory Investigational New Drug (EIND) study is designed to obtain preliminary imaging and fundamental biodistribution, metabolism and safety information to demonstrate early proof of concept. The information collected under this study will not be used for diagnostic purposes, to assess the subject's response to therapy, or for clinical management for the subject.

ELIGIBILITY:
Inclusion Criteria:

For Normal Volunteers

* Subject is ≥ 18 years old at the time of investigational product administration (Subject is male or female of any race / ethnicity)
* Subject or subject's legally acceptable representative provides informed consent
* Subject is capable of complying with study procedures
* Subject is capable of communicating with study personnel

For Cancer Subjects (same first four bullets as 'normals')

* Subject must have had a diagnostic imaging study and is suspected of having a primary or metastatic tumor(s) ( > 2 cm, except breast tumor)-sarcoma; melanoma; lung cancer [including small cell and non-small cell lung cancer (NSCL)]; high grade glioma (including glioblastoma multi-forms), anaplastic astrocytoma, and anaplastic oligodendroglioma; breast carcinomas, and head and neck tumors, including laryngeal squamous cell carcinoma
* Subject is scheduled to have a clinical [F-18]FDG PET scan within ± 7 days (with no interventions between the two PET scans) of the investigational, [F-18]RGD-K5 PET scan
* Subject is scheduled to undergo resection or biopsy of the target tumor as a result of routine clinical treatment
* Subject has not received any anti-angiogenic agents (e.g. bevacizumab, sorafenib, sunitinib) within 10 days prior to PET/CT imaging
* Subject has laboratory test results within the following ranges:
* AST(SGOT)/ALT(SGPT) ≤ 2.5 x institutional upper limits of normal
* Serum creatinine ≤ 1.5 institutional upper limits of normal
* Platelet count of > 75,000x106/L
* Hemoglobin value of > 9 g/dL
* ANC > 1.2 x 106 /mL

Exclusion Criteria 'Normals':

* Subject is < 18 at the time of investigational product administration
* Female subject is pregnant or nursing:
* by testing on site at the institution (serum or urine ßHCG) within 24 hours prior to the investigational product administration
* Subject is unable to remain still for duration of imaging procedure
* Subject has a history of renal disease
* Subject has previously received [F-18]RGD-K5 at any time, or any other investigational product in the past 30 days or will receive any other investigational product within 48 hours after the [F-18]RGD-K5 injection
* Subject has not been involved in an investigative, radioactive research procedure or therapeutic procedure within the past 6 months
* Subject has any other condition or personal circumstance including severe claustrophobia, severe dyspnea, severe back pain etc, that, in the judgment of the investigator, might interfere with the collection of complete good quality data
* Subject has a history of significant prescription or non-prescription drug, or alcohol abuse, including but not limited to marijuana, cocaine, heroin or derivatives.

For Cancer Subjects (first three bullets the same as 'normals')

* Subject is < 18 at the time of investigational product administration
* Female subject is pregnant or nursing:
* by testing on site at the institution (serum or urine ßHCG)
* Subject is unable to remain still for duration of imaging procedure
* Subject has known hyper or hypo-coagulation syndromes. (e.g., Protein C, S deficiency, Hemophilia A/B/C, Factor-V Leiden, etc.)
* Subject has previously received [F-18]RGD-K5 at any time, or any other investigational product in the past 30 days or will receive any other investigational product within 48 hours after the [F-18]RGD-K5 injection.
* Subject has inadequate tumor size (< 2 cm , except for breast tumor) or volume to allow for biopsy
* Subject has any other condition or personal circumstance including severe claustrophobia, severe dyspnea, severe back pain etc, that, in the judgment of the investigator, might interfere with the collection of complete good quality data
* Subject has a history of significant prescription or non-prescription drug, or alcohol abuse, including but not limited to marijuana, cocaine, heroin or derivatives.

Min Age: 18 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 16 (Estimated)
Dates: Start 2008-08; Primary Completion 2009-01 (Actual); Study Completion 2009-01 (Actual)

PRIMARY OUTCOMES:
To collect bio-distribution data to calculate dosimetry values in normals and obtain and evaluate PET images in cancer subjects for resolution of [F-18]RGD-K5 | imaging study-participation only days

CONTACTS AND LOCATIONS:
Overall Officials: Michael Yu, MD, Principal Investigator — Fox Chase Cancer Center, Dept of Nuclear Medicine, 333 Cottman Ave, Phila, PA 19111
Locations (1):
- Fox Chase Cancer Center, Philadelphia, Pennsylvania, United States

REFERENCES:
- [Derived] Doss M, Kolb HC, Zhang JJ, Belanger MJ, Stubbs JB, Stabin MG, Hostetler ED, Alpaugh RK, von Mehren M, Walsh JC, Haka M, Mocharla VP, Yu JQ. Biodistribution and radiation dosimetry of the integrin marker 18F-RGD-K5 determined from whole-body PET/CT in monkeys and humans. J Nucl Med. 2012 May;53(5):787-95. doi: 10.2967/jnumed.111.088955. Epub 2012 Apr 12. PMID 22499613